CLINICAL TRIAL: NCT01447615
Title: Bridges to the Future: Economic Empowerment for AIDS-Orphaned Children in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, PhD, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAA11950; 1R01HD070727-01 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Poverty; Orphaned Children; AIDS Orphans
Keywords: Orphaned children and youth; Economic empowerment; Uganda; HIV/AIDS; Sub-Saharan Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bridges (Experimental)
  Interventions: Behavioral: Bridges; Other: Usual Care
- Bridges PLUS (Experimental)
  Interventions: Behavioral: Bridges PLUS; Other: Usual Care
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Bridges — Each child participant in the Bridges Arm will receive the usual care in addition to a Child Development Account (CDA) to be used for secondary education by the AIDS-orphaned child. The CDA will be a matched savings account held in the child's name in a financial institution registered by the Central Bank (Bank of Uganda). The account will be matched with money from the program at a match rate of 1:1. Additionally, participants will receive: 1) twelve 1-2 hour workshops focused on asset building, future planning, and protection from risks; 2) mentorship sessions to reinforce learning and build optimism; and 3) a family income-generating /micro-enterprise promotion component for children enrolled in Bridges and their families.
  Other Names: Child Development Account
  Arms: Bridges
Behavioral: Bridges PLUS — Each child participant in the Bridges PLUS Arm will receive the usual care in addition to a Child Development Account (CDA) to be used for secondary education by the AIDS-orphaned child. The CDA will be a matched savings account held in the child's name in a financial institution registered by the Central Bank (Bank of Uganda). The account will be matched with money from the program at a match rate of 2:1. Additionally, participants will receive: 1) twelve 1-2 hour workshops focused on asset building, future planning, and protection from risks; 2) mentorship sessions to reinforce learning and build optimism; and 3) a family income-generating /micro-enterprise promotion component for children enrolled in Bridges PLUS and their families.
  Other Names: Child Development Account
  Arms: Bridges PLUS
Other: Usual Care — Participants in the usual care condition will receive usual care for AIDS-orphaned children in the study area. This includes: counseling, school lunches, and scholastic materials (textbooks and notebooks). Counseling will be provided by priests in the community (as is currently done).
  Other Names: Usual Services

SUMMARY:
Bridges to the Future: Economic Empowerment for AIDS-Orphaned Children in Uganda, represents the first study that measures medium-term efficacy and cost-effectiveness of a family economic empowerment intervention for AIDS-orphaned children. The usual care provided to AIDS orphans in sub-Saharan Africa consists mainly of informal counseling as well as limited material support (e.g., specifically school lunches, textbooks for the required subjects, and note-books). Given the challenges facing these children and their caregivers, further supports are needed in order to help them successfully make the transition from primary school to secondary school and into adolescence. In the context of resource-poor countries, interventions that improve families' economic capabilities are likely to be particularly consequential. Both theory and prior research indicate that economic instability (including poverty) constitutes one of the primary risk factors for AIDS-orphaned children's risk-taking behaviors (including sexual risk-taking), poor mental health functioning, and poor educational outcomes. Thus, the lack of economic security constitutes an important risk factor for AIDS-orphaned children. Yet, to-date, few interventions aimed at care and support of AIDS-orphaned children have incorporated components to address family-level poverty/economic instability of the children and their caregiving families. Within this context, there is a need for innovative interventions that promote sustainable (more than short-term) economic and behavior change among AIDS-orphaned children and create the supports necessary to sustain these changes.

DETAILED DESCRIPTION:
The overall goal of the proposed research is to evaluate the efficacy and cost-effectiveness of an innovative family-based economic empowerment intervention for AIDS-orphaned children. This will be accomplished via a three-group cluster randomized control trial (RCT). The three groups are: Bridges, Bridges PLUS, and usual care for AIDS-orphaned children. There will be five assessment points: baseline (pretest), 12, 24, 36, and 48-months post-intervention initiation.

The intervention, "Bridges to the Future" (Bridges) will be guided by asset-theory and both Bridges and Bridges PLUS will include the following intervention components tested in the two earlier pilot studies, SEED-Uganda and SUUBI-Uganda: 1) workshops focused on asset building, future planning, and protection from risks; 2) mentors to reinforce learning and build optimism; 3) a Child Development Account (CDA) that can be used for secondary education by the AIDS-orphaned child; and 4) a family income generating/micro-enterprise promotion component for children enrolled in Bridges and Bridges PLUS, and their families.

ELIGIBILITY:
Inclusion Criteria:

* An HIV/AIDS-orphaned child (a child who has lost one or both parents to HIV/AIDS)
* Enrolled in grade 5 or 6 of primary school
* Living within a family

Exclusion Criteria:

* Any child who does not self-identify as an HIV/AIDS-orphan
* Any child who is not enrolled in grade 5 or 6 of primary school
* Any child who is not living within a family at the time of enrollment

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1410 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Savings and Asset Accumulation | 12-month post-intervention follow-up assessment
  Increased confidence in saving ability and stronger financial stability. Accumulation of formal and informal savings and wealth/assets (e.g. livestock, type of housing, land); and change in attitudes toward saving.
Educational Achievement | 12-month post-intervention follow-up assessment
  School enrollment and attendance. Educational attainment, plans, and aspirations. Performance on National Primary Leaving Examinations.
Mental Health Functioning | 12-month post-intervention follow-up assessment
  Degree of hopefulness about the future. Ability to identify specific future goals. Level of mental health functioning. Depressive symptoms.
Sexual Risk-Taking Behavior | 12-month post-intervention follow-up assessment
  Ability to negotiate safe sex practices. Decreased intentions to engage in sexual risk behavior. Knowledge about and attitude toward HIV/AIDS and other STDs.
Savings and Asset Accumulation | 24-month post-intervention follow-up assessment
  Increased confidence in saving ability and stronger financial stability. Accumulation of formal and informal savings and wealth/assets (e.g. livestock, type of housing, land); and change in attitudes toward saving.
Educational Achievement | 24-month post-intervention follow-up assessment
  School enrollment and attendance. Educational attainment, plans, and aspirations. Performance on National Primary Leaving Examinations.
Mental Health Functioning | 24-month post-intervention follow-up assessment
  Degree of hopefulness about the future. Ability to identify specific future goals. Level of mental health functioning. Depressive symptoms.
Sexual Risk-Taking Behavior | 24-month post-intervention follow-up assessment
  Ability to negotiate safe sex practices. Decreased intentions to engage in sexual risk behavior. Knowledge about and attitude toward HIV/AIDS and other STDs.
Savings and Asset Accumulation | 36-month post-intervention follow-up assessment
  Increased confidence in saving ability and stronger financial stability. Accumulation of formal and informal savings and wealth/assets (e.g. livestock, type of housing, land); and change in attitudes toward saving.
Educational Achievement | 36-month post-intervention follow-up assessment
  School enrollment and attendance. Educational attainment, plans, and aspirations. Performance on National Primary Leaving Examinations.
Mental Health Functioning | 36-month post-intervention follow-up assessment
  Degree of hopefulness about the future. Ability to identify specific future goals. Level of mental health functioning. Depressive symptoms.
Sexual Risk-Taking Behavior | 36-month post-intervention follow-up assessment
  Ability to negotiate safe sex practices. Decreased intentions to engage in sexual risk behavior. Knowledge about and attitude toward HIV/AIDS and other STDs.
Savings and Asset Accumulation | 48-month post-intervention follow-up assessment
  Increased confidence in saving ability and stronger financial stability. Accumulation of formal and informal savings and wealth/assets (e.g. livestock, type of housing, land); and change in attitudes toward saving.
Educational Achievement | 48-month post-intervention follow-up assessment
  School enrollment and attendance. Educational attainment, plans, and aspirations. Performance on National Primary Leaving Examinations.
Mental Health Functioning | 48-month post-intervention follow-up assessment
  Degree of hopefulness about the future. Ability to identify specific future goals. Level of mental health functioning. Depressive symptoms.
Sexual Risk-Taking Behavior | 48-month post-intervention follow-up assessment
  Ability to negotiate safe sex practices. Decreased intentions to engage in sexual risk behavior. Knowledge about and attitude toward HIV/AIDS and other STDs.

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Ssewamala, PhD, Principal Investigator — Columbia University
Locations (1):
- International Center for Child Health and Asset Development, Masaka, Rakai and Masaka Districts, Uganda

REFERENCES:
- [Derived] Nabayinda J, Kizito S, Nabunya P, Namuyaba OI, Ssentumbwe V, Bahar OS, Torstein N, McKay M, Ssewamala FM. The Impact of an Economic Empowerment Intervention on Economic Security among AIDS-Orphaned Adolescents in Southern Uganda: the Moderating Role of Depression. AIDS Behav. 2026 Jan;30(1):242-252. doi: 10.1007/s10461-025-04862-0. Epub 2025 Aug 14. PMID 40810883
- [Derived] Ssewamala FM, Shu-Huah Wang J, Brathwaite R, Sun S, Mayo-Wilson LJ, Neilands TB, Brooks-Gunn J. Impact of a Family Economic Intervention (Bridges) on Health Functioning of Adolescents Orphaned by HIV/AIDS: A 5-Year (2012-2017) Cluster Randomized Controlled Trial in Uganda. Am J Public Health. 2021 Mar;111(3):504-513. doi: 10.2105/AJPH.2020.306044. Epub 2021 Jan 21. PMID 33476237
- [Derived] Nabunya P, Padgett D, Ssewamala FM, Courtney ME, Neilands T. Examining the nonkin support networks of orphaned adolescents participating in a family-based economic-strengthening intervention in Uganda. J Community Psychol. 2019 Apr;47(3):579-593. doi: 10.1002/jcop.22139. Epub 2018 Nov 5. PMID 30394541